CLINICAL TRIAL: NCT03202108
Title: A Feasibility Study to Evaluate the Acceptability of Krio, a Food for Special Medical Purposes (FSMP) for Use in the Ketogenic Diet (KD) With Regard to Product Tolerance, Compliance and Acceptability
Brief Title: Evaluation of Krio in Children and Adults With Epilepsy
Acronym: Krio
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Product manufacturing issues.
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-KRIO-2015-01-06
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Ketogenic Dieting; Epilepsy; Glucose Transporter Type 1 Deficiency Syndrome
Keywords: Ketogenic; Diet; Epilepsy; Glut-1 DS; Krio
MeSH Terms: conditions — Epilepsy; Glut1 Deficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consumption of Krio (Experimental): Incorporation of Krio into the daily diet.
  Interventions: Dietary Supplement: Krio

INTERVENTIONS:
Dietary Supplement: Krio — Krio is a ready to eat, chocolate-flavoured, solid bar containing 20g fat per 28g bar. It contains protein and carbohydrate with added sweetener and flavourings. It does not contain any added micronutrients. Krio is not for use as a sole source of nutrition.
  It has a fat to protein and carbohydrate ratio of 3 to 1, making it suitable for use in all versions of the ketogenic diet.
  This product is to be consumed daily under the direction of a dietitian.

SUMMARY:
Acceptability study to evaluate the gastrointestinal tolerance, palatability and participant compliance, over a 7-day period, of Krio for the dietary management of participants with intractable epilepsy or Glut-1 deficiency syndrome patients on a ketogenic diet.

DETAILED DESCRIPTION:
This is a prospective, acceptability study in fifteen (15) participants aged three (3) years and over, who are established on a ketogenic diet (KD), of Krio to aid in the management of their diet.

Participants will be provided with a 7-day supply of Krio and will be asked to complete a daily diary and short questionnaire to record information allowing assessment the following:

* Gastrointestinal tolerance
* Palatability
* Compliance

Krio is a Food for Special Medical Purposes (FSMP) and is intended for use in the KD. It has a fat to protein and carbohydrate ratio of 3 to 1. This makes it appropriate for inclusion in all versions of the KD: classical, medium chain triglyceride (MCT), modified Atkins diet (MAD) and low glycaemic index (LGI). It is suitable from 3 years of age.

Krio is presented as a ready to eat solid bar (28g), with no additional preparation required. It contains fat (20g per bar), protein and carbohydrate with added sweetener and flavourings. It does not contain any added micronutrients.

The recommended intake of the product for each participant will be determined by a dietitian. The quantity to be consumed daily will be recommended on an individual patient basis, but will be a minimum of 1 bar.

Product acceptability data from 15 participants are required in order to submit an application to the Advisory Committee on Borderline Substances (ACBS) for product registration.

ELIGIBILITY:
Inclusion Criteria:

i) Confirmed diagnosis of a condition requiring a KD, e.g. intractable epilepsy, Glut-1 DS.

ii) Aged three (3) years and over.

iii) Currently established on a KD for at least three (3) months, taken orally.

iv) Participant (or parent/guardian) considered by PI and dietitian to be fully proficient at managing the KD, and able to do this competently and accurately.

v) Participant (or parent/guardian) considered by PI and dietitian to be able to follow the protocol requirements and complete the diary and questionnaire.

vi) Freely given, written, informed consent from patient or parent/guardian.

vii) Freely given, written assent (if appropriate).

Exclusion Criteria:

i) Inability to comply with the study protocol, in the opinion of the investigator.

ii) Inability to comply with the ketogenic diet.

iii) Women who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study period.

N.B.: Women who become pregnant unexpectedly during this study may, in consultation with their doctor, continue on the study's dietary product if they wish but will not have any investigations that would not normally be carried out during pregnancy.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Product compliance daily diary | Days 1-7
  Quantitative assessments from subject questionnaires that allow evaluation of compliance with the study product, i.e. actual versus prescribed intake.
GI tolerance daily diary | Days 1-7
  Qualitative assessments from subject questionnaires that allow evaluation of the gastro-intestinal tolerance of the study product.
Ease of use questionnaire | Day 8
  Qualitative assessment from subject questionnaire that allows evaluation of the ease of use of the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Meskell, Principal Investigator — Leeds Teaching Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No